CLINICAL TRIAL: NCT01270152
Title: Determining the Safe Dosage of Ascorbic Acid Used in the Treatment of Occluded Totally Implanted Central Venous Catheter.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Christiane Inocencio Vasques, University of São Paulo, College of Nursing at Ribeirão Preto
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0925-0586
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Occluded Totally Implanted Central Venous Catheter
Keywords: ascorbic acid; catheterization central venous; nursing care
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group 50 mg ascorbic acid (Experimental): this arm received a dose of 50 mg of ascorbic acid administered inside the catheter and maintained for up to 60 minutes
  Interventions: Drug: Ascorbic Acid
- group 100mg ascorbic acid (Experimental): this arm received a dose of 100 mg of ascorbic acid administered inside the catheter and maintained for up to 60 minutes
  Interventions: Drug: Ascorbic Acid
- group 200mg ascorbic acid (Experimental): this arm received a dose of 200 mg of ascorbic acid administered inside the catheter and maintained for up to 60 minutes
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — comparing three different doses of ascorbic acid: 50 mg, 100 mg and 200 mg administered inside the catheter and maintained for up to 60 minutes
  Other Names: Ascorbic Acid to restore catheter patency

SUMMARY:
The hypothesis of the study is to evaluate whether ascorbic acid is able to clear totally implanted central venous catheter

DETAILED DESCRIPTION:
Totally implanted catheter is often occluded and thrombolytic drugs are usually used to restore permeability. In Brazil, the ascorbic acid has been used successfully by a service specialist in cancer treatment. However, no literature on international research that evaluates the efficacy and safety of this procedure. That was why it was decided to develop this research.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of partial or complete obstruction of the totally implanted central venous catheter;
* No signs of inflammation in the area of the port.

Exclusion Criteria:

* Use of oral anticoagulants or intravenous administration in the last seven days;
* Diagnostic and / or suspected infection in the totally implanted central venous catheter;
* Rupture, displacement or fissure of the totally implanted central venous catheter;
* Presence of thrombosis in the vein where the catheter is inserted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Restore patency | 60 minutes after administration of ascorbic acid
  the ascorbic acid is administered and remains inside the catheter within 60 minutes. The recovery of permeability is checked every 15 minutes until the maximum of 60 minutes

SECONDARY OUTCOMES:
Eosinophil count | within 24 hours
  the count of eosinophils was determined by collecting blood sample immediately prior to administration of ascorbic acid and 24 hours after

CONTACTS AND LOCATIONS:
Overall Officials: Christiane I Vasques, Doc, Principal Investigator — University of São Paulo, College of Nursing at Ribeirão Preto
Locations (1):
- Clinical Hospital of Medicine College of Ribeirão Preto, University of São Paulo, Ribeirão Preto, São Paulo, Brazil